CLINICAL TRIAL: NCT02652806
Title: A Phase 3, Randomized, Open-Label, Active-Controlled Study of Efficacy and Safety of FG-4592 for Treatment of Anemia in Subjects With Chronic Kidney Disease on Dialysis
Brief Title: FG-4592 for Treatment of Anemia in Subjects With Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-806
Record Dates: First submitted 2015-12-31; First posted 2016-01-12 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-02

CONDITIONS: Anemia
Keywords: Chronic Kidney Disease
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — roxadustat; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FG-4592 (Experimental): Intervention is investigational treatment FG-4592
  Interventions: Drug: FG-4592
- EPO (Active Comparator): Intervention is subject's current dose of Li Xue Bao (epoetin alfa)
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: FG-4592
  Arms: FG-4592
Drug: Epoetin Alfa
  Other Names: Li Xue Bao
  Arms: EPO

SUMMARY:
This is a randomized, multicenter, open-label, active-controlled study of the treatment of anemia in subjects with CKD on dialysis, with treatment up to 52 weeks.

DETAILED DESCRIPTION:
This is a randomized, multicenter, open-label, active-controlled study of the treatment of anemia in subjects with CKD on dialysis. Eligible subjects are randomized to FG-4592 or epoetin alfa at a ratio of 2:1. The primary endpoint is Hb mean change from baseline averaged over Weeks 23 to 27.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 75 years
2. Subject has voluntarily signed and dated an informed consent form (ICF), approved by an Ethics Committee (EC), after the nature of the study has been explained and the subject has had the opportunity to ask questions; a separate ICF is needed for subjects participating in the PK Sub-study.
3. "Chronic kidney disease with end-stage renal disease (ESRD) on either adequate hemodialysis (HD) or adequate peritoneal dialysis for a minimum of 16 weeks prior to Day 1: For subjects undergoing HD, the vascular access must be via native arteriovenous (AV) fistula or graft, or permanent, tunneled catheter."
4. Subjects must be on stable doses of IV or subcutaneous (SC) injections of epoetin alfa for at least 6 weeks prior to Day 1 (average dose ≤15,000 IU/week)
5. Mean of the two most recent central laboratory Hb values during the Screening Period, obtained at least 6 days apart, must be 9.0 g/dL to 12.0 g/dL, inclusive, with a difference of \≤1.5 g/dL between the highest and the lowest Hb values.
6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 x upper limit of normal (ULN), and normal total bilirubin at screening visit except for subjects with Gilberts syndrome (based on central laboratory results).
7. Body weight: 45 to 100 kg inclusive 8 Subjects agree not to start taking any new Traditional Chinese Medicine (TCM) for anemia and not to change dose, schedule, or brand of any prescreening TCM for anemia from beginning of Screening Period through end of Follow-up Period.

Exclusion Criteria:

1. Any clinically significant infection or evidence of an active underlying infection.
2. Positive for any of the following: human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus antibody (anti-HCV Ab).
3. Chronic liver disease.
4. New York Heart Association Class III or IV congestive heart failure.
5. Myocardial infarction, acute coronary syndrome, stroke, seizure, or a thromboembolic event (eg, deep venous thrombosis or pulmonary embolism) within 52 weeks prior to Day 1.
6. Uncontrolled hypertension in the opinion of the investigator (eg, that requires change in anti-hypertensive medication within 2 weeks prior to randomization).
7. Diagnosis or suspicion (eg, complex kidney cyst of Bosniak Category II or higher) of renal cell carcinoma as shown on screening renal ultrasound.
8. History of malignancy except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, or in situ cancer at any site.
9. Chronic inflammatory disease other than glomerulonephritis that could impact erythropoiesis (eg, systemic lupus erythematosis [SLE], rheumatoid arthritis, celiac disease).
10. Clinically significant gastrointestinal bleeding.
11. Known history of myelodysplastic syndrome, multiple myeloma, hereditary hematologic disease such as thalassemia, sickle cell anemia, pure red cell aplasia, or other known causes for anemia other than CKD, hemosiderosis, hemochromatosis, known coagulation disorder, or hypercoagulable condition.
12. Any prior functioning organ transplant or a scheduled organ transplantation, or anephric.
13. Anticipated elective surgery that could lead to significant blood loss during the study period.
14. Anticipated use of dapsone or acetaminophen (paracetamol) >2.0 g/day, or >500 mg per dose repeated every 6 hours for more than 3 days.
15. Serum albumin <2.5 g/dL.
16. Androgen, deferoxamine, deferiprone, or deferasirox therapy within 12 weeks prior to Day 1.
17. Life expectancy of <12 months.
18. Blood transfusion within 12 weeks prior to Day 1 or anticipated need for transfusion.
19. IV iron supplement during the Screening Period and /or unwilling to withhold IV iron.
20. Immune suppressive or systematic steroid treatment within 12 weeks prior to Day 1.
21. History of alcohol or drug abuse within the past 2 years and inability to avoid consumption of more than >3 alcoholic beverages per day.
22. Prior treatment with FG-4592 or any hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI).
23. Use of an investigational medication or treatment, participation in an investigational interventional study, or carryover effect of an investigational treatment expected during the study.
24. Women who are pregnant or breastfeeding.
25. Women of childbearing potential and men with sexual partners of child bearing potential who are not using adequate contraception.
26. Any medical condition that, in the opinion of the investigator, may pose a safety risk to a subject in this study, may confound efficacy or safety assessment, or may interfere with study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01-24 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Hb mean change from baseline | Weeks 23 to 27.
  Hb mean change from baseline

SECONDARY OUTCOMES:
Mean change from baseline in low-density lipoprotein (LDL) cholesterol | Weeks 25-27
  Mean change from baseline in low-density lipoprotein (LDL) cholesterol
Number of subjects with a Hb response | Weeks 23-27
  Number of subjects with a Hb response (as defined per protocol)
Percent of subjects with a Hb response | Weeks 23-27
  Percent of subjects with a Hb response (as defined per protocol)
Effect on iron metabolism | Week 27
  Measurement of serum iron
Proportion of subjects with exacerbation of hypertension | Up to Week 27
  Proportion of subjects with exacerbation of hypertension, meeting at least one of the following criteria up to Week 27:
  * Increase in anti-hypertensive medication use,
  * Adverse event of hypertension, or
  * Increases from baseline in blood pressure confirmed by repeat measurement at next visit unless anti-hypertensive medications are changed.
Mean change from baseline in predialysis and postdialysis mean arterial blood pressure | Weeks 23-27
  Mean arterial blood pressure measured pre-and post-dialysis.
Number of subjects with treatment-emergent adverse events (TEAEs). | Week 1 to up to Week 53
  Number of subjects with treatment-emergent adverse events (TEAEs).
Percent of subjects with treatment-emergent adverse events (TEAEs). | Week 1 to up to Week 53
  Percent of subjects with treatment-emergent adverse events (TEAEs).
Changes from baseline in vital signs | Week 1 to up to Week 53
  Measurement of vital signs
Changes from baseline in ECG findings. | Week 1 to up to Week 53
  ECG recordings.
Changes from baseline in clinical laboratory values. | Week 1 to up to Week 53
  Clinical laboratory values.
Number and % of subjects on rescue therapy during study treatment. | Week 1 to up to Week 53
  Number and % of subjects on rescue therapy during study treatment.
Time to rescue therapy from date of first dose during study treatment. | Week 1 to up to Week 53
  Time to rescue therapy from date of first dose during study treatment.

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - 301 Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Pekingg University, People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated hospital of Third Military Medical University (Southwest Hospital), Chongqing, Chongqing Municipality
  - Lan Zhou University Second Hospital, Lanzhou, Gansu
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Affiliated hospital of Guangxi Medical University, Nanning, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Hospital of Baotou Medical School of Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medication, Shanghai, Shanghai Municipality
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medication, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan Universtiy, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Chen N, Hao C, Liu BC, Lin H, Wang C, Xing C, Liang X, Jiang G, Liu Z, Li X, Zuo L, Luo L, Wang J, Zhao MH, Liu Z, Cai GY, Hao L, Leong R, Wang C, Liu C, Neff T, Szczech L, Yu KP. Roxadustat Treatment for Anemia in Patients Undergoing Long-Term Dialysis. N Engl J Med. 2019 Sep 12;381(11):1011-1022. doi: 10.1056/NEJMoa1901713. Epub 2019 Jul 24. PMID 31340116